CLINICAL TRIAL: NCT05424289
Title: The Predictive Value of Videoryngoscopy in Preoperative Airway Evaluation in Obese Patients
Status: Completed | Type: Observational
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, derya özkan, Professor MD, Diskapi Teaching and Research Hospital
Other Study IDs: SBU 2022
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Difficult Intubation in Obesity
Keywords: difficult airway prediction, videolaryngoscopy, obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes

INTERVENTIONS:
Device: videolaryngoscope — Videolaryngoscope is a high-resolution micro camera mounted on the tip of a curved blade connected to small portable digital monitor improves the view of the vocal cords

SUMMARY:
The aim of this study is the evaluation of preoperativevideolaryngoscopy, as a possible predictor of difficult laryngoscopy and intubation during elective general anesthesia in an obese population.

Videolaryngoscopy is a minimally invasive examination performed during difficult intubation evaluation but not used routinely . On the other hand, current strategies used to predict the ease of intubation are still not sufficiently sensitive and specific. An unexpected difficult or failed intubation at the induction of general anesthesia is a seriuos, and potentially fatal, emergency in anesthesia.

In literature, a correlation between anatomical and functional parameters highlighted by videolaryngoscopy and difficulty of laryngoscopy and intubation has never been demonstrated nor indagated. There is only some case reports related evaluation of diffucult airway by videolaryngoscopy .

If proven, this might give the Anesthestiologist further information about the expected difficulty of laryngoscopy and intubation, guiding a different anesthesiological strategy.

DETAILED DESCRIPTION:
This is a prospective, single-center, observational study. Aim of this study is the evaluation of preoperative videolaryngoscopy as a predictor of difficult laryngoscopy and intubation during elective general anesthesia in an obese population. Unexpected difficult of failed intubation is a serious, and potentially fatal, occurrence at the induction of general anesthesia. However, current strategies used to predict the ease of intubation are still not sufficiently sensitive and specific.

Routine airway evaluation will be performed by the same anesthesiologist for patients with a BMI above 30 who will undergo general anesthesia for scheduled surgery. In the preoperative operating room, these patients will undergo videoingoscopy and a POGO score will be applied (10% lidocaine will be sprayed on tonsil sites).

The investigators who do not performed preoperative videolaryngoscopy evaluation will be also collected data about the preoperative evaluation made by the Anesthesiologist as well as the effective difficulty of laryngoscopy and intubation encountered at the induction of general anaesthesia, expressed by the Cormack - Lehane scale and the Intubation Difficulty Scale (IDS) as described in literature.

General anesthesia will be performed as usual and will not be influenced by videolaryngoscopic evaluation as the Anesthesiologist will be blind to it, and he/she will be free to choose the best anesthesiological plan for his/her patient; whether an elective awake intubation will be chosen, this will exclude the patient from the study.

For safety reasons, the only exception to blindness is an expected difficulty of intubation (POGO score 0%) by senior anesthesiologist, based upon the physician's experience. In this case, he will talk to the Anesthesiologist about and the patient will be excluded from the study.

Preoperative data obtained by videolaryngoscopy and intraoperative data recorded by the Anesthesiologist will be matched and analyzed, to explore a possibile relationship.

ELIGIBILITY:
Inclusion Criteria:

* Candidate to elective surgery under general anesthesia Body mass index (BMI) 30<

Exclusion Criteria:

* Subjects with suspect or ascertained malignancy of the nose, mouth, phayrx, or larynx that may interfere with tracheal intubation Subjects with tracheostomy Subjects candidate to elective awake intubation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Candidate to elective surgery under general anesthesia obese patients BMI 30<
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Difficulty of tracheal videolaryngoscopy | Intraoperative (single assessment)
  The difficulty of tracheal laryngoscopy is described with the modified Cormack - Lehane Scale.

SECONDARY OUTCOMES:
Difficulty of tracheal intubation | Intraoperative (single assessment)
  The difficulty of intubation is described with and the Intubation Difficulty Scale (IDS)

CONTACTS AND LOCATIONS:
Locations (1):
- Ministry of Health Diskapi Yildirim Beyazit Research and Training Hospital departement of 1. Anesthesiology, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Utada S, Okano H, Miyazaki H, Niida S, Horiuchi H, Suzuki N, Otsuka T, Furuya R. Awake intubation with videolaryngoscopy and fiberoptic bronchoscope. Clin Case Rep. 2022 Jan 11;10(1):e05274. doi: 10.1002/ccr3.5274. eCollection 2022 Jan. PMID 35035964
- [Result] Heinrich S, Birkholz T, Irouschek A, Ackermann A, Schmidt J. Incidences and predictors of difficult laryngoscopy in adult patients undergoing general anesthesia : a single-center analysis of 102,305 cases. J Anesth. 2013 Dec;27(6):815-21. doi: 10.1007/s00540-013-1650-4. Epub 2013 Jun 9. PMID 23748552
- [Result] Cormack RS, Lehane J. Difficult tracheal intubation in obstetrics. Anaesthesia. 1984 Nov;39(11):1105-11. PMID 6507827
- [Result] Adnet F, Borron SW, Racine SX, Clemessy JL, Fournier JL, Plaisance P, Lapandry C. The intubation difficulty scale (IDS): proposal and evaluation of a new score characterizing the complexity of endotracheal intubation. Anesthesiology. 1997 Dec;87(6):1290-7. doi: 10.1097/00000542-199712000-00005. PMID 9416711